CLINICAL TRIAL: NCT03184532
Title: Bedside Gastric Ultrasound for Assessment of ASA Preoperative Starving Guidelines Accuracy: Diabetic vs Non Diabetic Patients
Acronym: gastric US
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Healthpoint Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Elahl, anesthesia consultant, Healthpoint Hospital
Other Study IDs: rec003
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Evaluation of ASA Fasting Recommendations in Diabetic Patients
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- D: diabetic patients
  Interventions: Diagnostic Test: ultrasound
- ND: non-diabetic patients
  Interventions: Diagnostic Test: ultrasound

INTERVENTIONS:
Diagnostic Test: ultrasound — ultrasound examination of pyloric antrum

SUMMARY:
To reduce the risk of perioperative pulmonary aspiration of gastric contents, oral intake of liquids or solids is not allowed for certain periods. Recently, the ultrasound (US) is used to evaluate the volume and the nature of the stomach content. In its latest recommendations, the American Society of Anesthesiologists (ASA) shortened the duration preoperative fasting. The aim of the study is to evaluate the efficacy of ASA recommendations in diabetic patients using ultrasound (US) scanning of the stomach (antrum).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective orthopedic procedures.

Exclusion Criteria:

* Patients with BMI > 35 kg.m-2, age <18y, ASA physical state >II, fasting more than 6hs, or with gastric diseases will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective orthopedic procedures.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2017-12-15 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
gastric volume | bedside test 5 minutes